CLINICAL TRIAL: NCT02782910
Title: Smartphone-based Ambulatory Assessment of Early Warning Signs, Including Personalized Real-time Data-driven Therapeutic Interventions, in the Long-term Treatment of Bipolar Disorders.
Brief Title: Smartphone-based Ambulatory Assessment of Early Warning Signs
Acronym: BipoLife_A3
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Technische Universität Dresden (Other)
Collaborators: German Federal Ministry of Education and Research (Other Government); KIT (Karlsruher Institut für Technologie) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: BipoLife_A3
Record Dates: First submitted 2015-08-03; First posted 2016-05-25 (Estimated); Last update posted 2018-05-29 (Actual); Status verified 2018-05

CONDITIONS: Bipolar Disorder
MeSH Terms: conditions — Bipolar Disorder

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- SBAA+ (Experimental): Upon exceeding pre defined SBAA-threshold limits during the randomisation phase the treating physician is alerted (+) to this signal and required to contact the patient so as to assess the current mental status and collaboratively discuss the potential need for medical/psychiatric treatment with the patient.
  Interventions: Device: Smartphone-Based Ambulatory Assessment, Feedback via physician
- SBAA (No Intervention): Continuous monitoring will occur analogous to SBAA+. Exceeding the pre defined SBAA-threshold will not result in any action taken.

INTERVENTIONS:
Device: Smartphone-Based Ambulatory Assessment, Feedback via physician — Participants in the experimental condition SBAA+ will be contacted by their treating physician, once the predefined threshold for Smartphone activity is exceeded.
  Other Names: Smartphone feedback via server
  Arms: SBAA+

SUMMARY:
Bipolar disorders are severe chronic disorders, marked by recurrent episodes of depression and (hypo)mania. The disorder usually emerges in early adulthood and tends to have a highly unpredictable course. Prevention of these episodes is essential, as they are associated with marked impairment in social and occupational functioning. The investigators propose to conduct a randomized, multi-center, observer-blind, parallel group controlled trial with an 78 week (18 month) intervention phase to test the hypothesis that continuous ambulatory real-time monitoring of early warning signs for new depressive or (hypo)manic episodes by smartphone based, innovative technology (e.g. GPS, acceleration sensor), including individual threshold- based early intervention for these early warning signs, will prolong time to a new mood episode and reduce hospitalizations (intervention group). In the control group ambulatory monitoring of early warning signs for emerging depressive or (hypo)manic episodes will occur in an identical manner, but the results will not be transmitted to the treating psychiatrist. All patients in this trial, irrespective of their group assignment, will receive guideline-based, state-of-the-art maintenance treatment.

DETAILED DESCRIPTION:
Symptomatic outpatients with bipolar disorders I/II , will be consecutively assessed for eligibility. After having signed informed consent patients will receive open, guideline-based, state-of-the-art treatment for their current symptomatology ((hypo)manic and/or depressed) for up to 16 weeks. As soon as patients meet stabilisation criteria (YMRS total score < 12 and IDS total score < 12) they will be equipped with a study smartphone, for exclusive use during the study period, to assess the parameters of interest (activity, communication pattern, sleep pattern) and define the individual symptoms' threshold during 4 consecutive weeks of stabilisation . If patients fulfil randomization criteria (4 consecutive weeks with YMRS total score < 12 and IDStotal score < 12), they will enter the observer (rater) - blind, intervention phase, which will continue for 18 months (78 weeks). At randomization patients will be assigned to either the Smartphone-Based Ambulatory Assessment group, including real-time data capture and data-driven, individual symptoms' threshold-defined therapeutic interventions (SBAA+), in addition to state-of-the-art maintenance treatment or the Smartphone-Based Ambulatory Assessment group, only including real-time data capture (SBAA), in addition to state-of-the-art maintenance treatment.

ELIGIBILITY:
Inclusion Criteria:

* Bipolar Disorders (I/II)

  * > 3 affective episodes in 5 years prior to index episode, with one of them being a (hypo)manic episode
  * Age > 18 years
  * Male or female
  * Inpatients or outpatients
  * Smartphone usage
  * Each patient must have a level of understanding sufficient to agree to all tasks required by the protocol.
  * Patients must be considered reliable.
  * Each patient must sign an informed consent document prior to enrollment.

Exclusion Criteria:

* Current substance use disorder (except for tobacco and caffeine), moderate or severe, at enrolment
* Borderline personality disorder, antisocial personality disorder
* Dementia, organic brain disorders
* Unstable/inadequately treated medical illness
* Clinically significant cardiac, renal, hepatic, neoplastic or cerebrovascular disease
* Any medical condition posing a significant risk regarding adherence to study protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2017-01-01 (Actual); Primary Completion 2020-07 (Estimated); Study Completion 2020-07 (Estimated)

PRIMARY OUTCOMES:
Time to relapse | Duration of trial after randomisation (total of 18 months)
  Time until new affective episode (hypomanic, manic, mixed, depressed) according to DSM V criteria

SECONDARY OUTCOMES:
Total time in episode | Duration of trial after randomisation (total of 18 months)
  Percentage of assessments during intervention phase at which the criteria for an affective episode are met
Severity of manic symptomatology | Duration of trial after randomisation (total of 18 months)
  Average severity of manic symptoms at assessments during intervention phase, as judged by YMRS score
Severity of depressive symptomatology | Duration of trial after randomisation (total of 18 months)
  Average severity of depressive symptoms at assessments during intervention phase, as judged by IDS score.
Total hospitalisation | Duration of trial after randomisation (total of 18 months)
  Percentage of assessments during intervention phase at which the patient was hospitalized for an affective episode

CONTACTS AND LOCATIONS:
Overall Officials: Michael Bauer, MD, Study Director — Technische Universität Dresden
Locations (1):
- Department of Psychiatry and Psychotherapy, Dresden, Saxony, Germany

REFERENCES:
- [Derived] Muhlbauer E, Bauer M, Ebner-Priemer U, Ritter P, Hill H, Beier F, Kleindienst N, Severus E. Effectiveness of smartphone-based ambulatory assessment (SBAA-BD) including a predicting system for upcoming episodes in the long-term treatment of patients with bipolar disorders: study protocol for a randomized controlled single-blind trial. BMC Psychiatry. 2018 Oct 26;18(1):349. doi: 10.1186/s12888-018-1929-y. PMID 30367608
- See also: Central study website — http://www.bipolife.org